CLINICAL TRIAL: NCT06370897
Title: A Prospective and Retrospective Observational Study of Symptoms and Mechanisms of Recovery in People With Inner Ear Decompression Sickness (IEDS)
Brief Title: Prediction & Mechanisms of Recovery Following IEDS
Status: Not yet recruiting | Type: Observational
Sponsor: University of Plymouth (Other)
Responsible Party: Principal Investigator, Jon Marsden, Professor of Rehabilitation, University of Plymouth
Other Study IDs: 337421
Record Dates: First submitted 2024-04-08; First posted 2024-04-17 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Decompression Sickness
Keywords: vestibular, inner ear
MeSH Terms: conditions — Decompression Sickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prospective Cohort: Divers admitted with suspected IEDS
- Retrospective Cohort: Divers diagnosed with Inner ear decompression sickness (IEDS) at Deep Diving Research Centre within past 10 years

SUMMARY:
Inner Ear Decompression sickness (IEDS) accounts for 20% of all types of decompression sickness (the bends) in divers. The condition commonly affects the peripheral vestibular system (inner ear). IEDS results in acute symptoms of dizzyness (vertigo) and imbalance. Even with the recommended treatment of hyperbaric oxygen therapy some people do not recovery fully. However, even in the presence of a permanent vestibular deficit many people can show a behavioural recovery where symptoms improve over time. Recovery can be aided by vestibular rehabilitation (VR) which is now routine for acute IEDS but was not provided before 2021, and is not widespread across the UK (United Kingdom) or world, meaning people may have a suboptimal recovery.

This project will investigate if and how people recover after an acute episode of IEDS and whether people who had IEDS in the past show changes in the central (brain) processing of vestibular function and in symptoms of dizziness, balance and posture.

This project has two main parts. Part one is a prospective observational study where people with an acute onset of IEDS are serially monitored while they are receiving hyperbaric treatment and VR over 10-14 days. Part two is a retrospective observational study where who have had IEDS in the past 15 years are re-assessed in a one-off session. The tests in both parts involve clinical tests and specialist eye movement recordings that assess vestibular function. We will also determine the site of any vestibular pathology by using selective stimulation of the vestibular end organ or nerve and assess whether there are any changes in how the structure and function of central vestibular pathways in the brain. In people with chronic IEDS with vestibular symptoms we will offer participants a course of VR over 12 weeks and assess whether this is associated with any improvement in symptoms.

DETAILED DESCRIPTION:
Decompression sickness after diving can occur following a rapid ascent. Here, nitrogen, absorbed by the body when breathing compressed air at depth, comes out of solution and forms microbubbles in the blood. Inner ear decompression sickness (IEDS) accounts for approximately 20% of all cases of decompression sickness. The vestibular system is involved in ~85% cases of IEDS resulting in symptoms of vertigo, nausea, vomiting and unsteadiness with hearing loss and tinnitus.

The strong association of IEDS with a patent foramen ovale (50-73% of cases) suggests that a shunted venous gas embolism causes damage to the vestibular apparatus, which is particularly vulnerable due to its low perfusion and thus slow inert gas washout, compared to the cochlea and other brain structures. It is hypothesised that the nitrogen bubbles within the blood vessels trigger an inflammatory reaction in the endothelium with a coagulation cascade that leads to hypoxic injury and/or that there is direct damage to the membranous labyrinth. Animal models of rapid decompression suggest that it can cause a haemorrhage within the labyrinth with ectopic bone growth and fibrosis occurring over the next month. Advances in the imaging of the inner ear using a gadolinium-based contrast agent (GBCA) allow us to explore structural changes in human divers. Imaging can also help to differentially diagnose another potential cause of diving induced dizziness, superior structural dehiscence syndrome

Decompression sickness and the subsequent inflammatory response requires emergency treatment using with hyperbaric oxygen. The effects of hyperbaric therapy and rehabilitation are not uniform across participants, factors affecting recovery include a high clinical score on admission and a delay in hyperbaric recompression of over 6 hours. Complete recovery is seen in only about 30% of cases. Previous studies have highlighted that people who do not fully recover can have a variety of symptoms that can affect work, hobbies and well-being. These include feelings of instability in some situations (working at a height and with movement) and imbalance in the dark or when changing position.

In people with permanent vestibular pathology, symptoms can still improve due to central adaptive processes within the brain termed vestibular compensation. Clinical studies in other types of peripheral vestibular dysfunction show that it is possible to facilitate the compensation process and symptom recovery through vestibular rehabilitation. Early access to vestibular rehabilitation is now routine practice at the Diving Diseases Research Centre (DDRC) where patients are treated in the South-West UK. This is coupled to diagnosis and monitoring of vestibular function using objective laboratory tests (rotary testing) and clinical tests.

Animal studies highlight the mechanisms underlying vestibular compensation following a peripheral nerve lesion. These focus on changes in the interconnections between brainstem nuclei (e.g. vestibular nuclei) and the cerebellum and re-weighting of the relative importance of multi-sensory sensory inputs. Human studies in chronic peripheral dysfunction also suggest there are recovery-related changes in cortical areas that normally process vestibular information over time. Functional changes in the acute stages include an increase in contralesional activity in the parietoinsular vestibular cortex as well as interlinked subcortical areas (posterolateral thalamus, anterior cingulate gyrus, pontomesencephalic brainstem, hippocampus) with a decrease in activity was seen in the visual, somatosensory and auditory cortices. Structural changes over the first 3 months post lesion include increases in grey matter volume in the vestibular cortex, bilateral hippocampus, visual cortices and the cerebellum.

Within the DDRC vestibular rehabilitation has only been routinely undertaken for people diagnosed with IEDS since 2021. As complete recovery is seen in only about 30% of cases [9]; this suggests that there may be a cohort of patients with residual vestibular symptoms. In surveys of the aural and vestibular effects of diving, including those conducted by the DDRC, 79% (of 790 respondents) have reported aural related problems after learning to dive. Of those with reported problems 46% did not seek any medical advice and 39% specifically reported dizziness / vertigo. In total this suggests that at least 14% of all divers may have undiagnosed vestibular problems that could benefit from vestibular rehabilitation. A case review highlights that since 1999 there have been 79 cases of clinically diagnosed IEDS at the DDRC. Therefore, there is a need to assess and provide rehabilitation support to people with past IEDS and potentially in the future a larger cohort of divers with previously undiagnosed symptoms.

This study plans to:

undertake a prospective observational study where people with acute onset IEDS are followed up. This will include the current battery of clinical and laboratory (rotary) tests but also additional optional clinical and physiological testing (Vestibular Evoked Myogenic Potentials VEMPs), imaging (Diffusor Tensor Imaging DTI and functional Magnetic Resonance Imaging f MRI) and semis-structured interviews in the acute (1-14 days) and chronic (3 months and 12 months) stage.

We will also:

undertake a retrospective cross-sectional study of people who have previously been managed for IEDS by the DDRC. Here we will undertake the same battery of tests as for the prospective study which includes measures of potential risk factors and patient reported outcome measures. We will also take this opportunity to explore people's symptoms post IEDS and their views on future rehabilitation trials. In those with remaining vestibular symptoms and signs we will provide advice on vestibular rehabilitation by qualified personnel with follow up as required. We will compare our data to a cohort of healthy controls of a similar age and gender distribution.

ELIGIBILITY:
Prospective Study :

Inclusion

• Divers admitted with suspected IEDS

Exclusion

* Medically unstable
* Unstable orthopaedic deficits

Retrospective study :

Inclusion

• Divers diagnosed with IEDS at DDRC within past 10 years

Exclusion

• We will include all co-morbidities as these could affect prognosis and recovery following IEDS.

Healthy control comparator group :

Normative data will be gathered on an age matched group. There will be at least 10 participants for each decade (<30yrs ,30-40yrs, 40-50 yrs,50-60yrs,60-70 yr.)

Inclusion criteria:

• Adults over 18 years

Exclusion criteria:

• Neurological, sensory or orthopaedic conditions that could affect balance.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population: Divers
  Exposure: Dive resulting in IEDS symptoms
Sampling Method: Non-Probability Sample
Enrollment: 41 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Side of peripheral vestibular damage: Prospective cohort | T0=baseline within 24 hours of IEDS in the prospective cohort
  Side (left or right) of vestibular dysfunction as determine by video head impulse test (v HIT) testing
Site of peripheral vestibular damage: Prospective cohort | T0=baseline within 24 hours of IEDS in the prospective cohort
  Site of dysfunction: semi-circular canals affected as determine by v HIT testing. One or a combination of Horizontal, anterior or posterior canals.
Extent of peripheral vestibular damage: Prospective cohort | T0=baseline within 24 hours of IEDS in the prospective cohort
  VOR gain (unit less) as measured by v HIT at T0 (Range 0-1 higher values are better outcome)
Side of peripheral vestibular damage: Retrospective cohort | 1 time point: 0-10 years post injury
  Side (left or right) of vestibular dysfunction as determine by video head impulse test (v HIT) testing
Site of peripheral vestibular damage:Retrospective cohort | 1 time point: 0-10 years post injury
  Site of dysfunction: semi-circular canals affected as determine by v HIT testing.One or a combination of Horizontal, anterior or posterior canals.
Extent of peripheral vestibular damage:Retrospective cohort | 1 time point: 0-10 years post injury
  VOR gain (unit less) at T0 (Range 0-1 higher values are better outcome)

SECONDARY OUTCOMES:
VOR gain v HIT: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in VOR gain assessed through V HIT test . Gain is unit less and range from 0-1 where higher values indicate a better clinical outcome.
VOR gain: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in VOR gain assessed through sinusoidal rotation in the dark . Gain is unit less and range from 0-1 where higher values indicate a better clinical outcome.
VOR Time constant:Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0)in VOR time constant in response to a step rotation (initial 140°/s acceleration/deceleration and a 60°/s fixed-chair velocity) stimulus . Time constant (seconds) where a higher time constant is clinically better. Range 0-40s.
Patient reported outcome measure: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in PROM (patient reported outcome measure) vertigo severity scale.15 questions rated 0-4. Score range =0-60 where lower scores indicate a better clinical outcome
Clinical measure of walking: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in Dynamic Gait Assessment (DGA). Eight tasks scored 0-3. Total range = 0-24 with a higher score indicating better walking ability.
Clinical measure of balance: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in Clinical measures of balance sharpened Romberg (tandem stance). The length of time a person is able to stand in the eyes open, tandem stance position is recorded up to a maximum of 30 seconds.
Posturography: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in Postural sway quotient. Postural sway (mm/s) is measured via force plates. The ratio of the sway with eyes open and eyes closed is calculated (unitless ratio).
Perception of verticality: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in Rod and Disk test: The ability to orientate a line to vertical is assessed with / without visual distractors. The error from vertical is recorded in degrees. Outcomes range from 0-180 degrees where lower numbers indicate better verical perception.
Functional MRI response to an optokinetic stimulus: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in Regions of interest will also assess changes in activation with an optokinetic stimulus compared to rest in cortical and subcortical sites that process vestibular information namely the insulo-parietal cortex and hippocampus and sites that process other sensory information namely the visual cortex and somatosensory cortex
Vestibular Evoked myogenic Potentials latency: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in Galvanic and Auditory Vestibular Evoked myogenic Potentials (VEMPs) will be assessed and the latency of evoked responses measured in milliseconds.
Vestibular Evoked myogenic Potentials amplitude: Prospective Study | 7-10 days , 3 months and 12 months post injury
  Change from baseline (T0) in Galvanic and Auditory Vestibular Evoked myogenic Potentials (VEMPs) will be assessed and the amplitude of evoked responses measured in millivolts.
VOR gain: Retrospective Study | 7-10 days , 3 months and 12 months post injury
  VOR gain assessed through sinusoidal rotation in the dark . Gain is unit less and range from 0-1 where higher values indicate a better clinical outcome.
VOR Time constant: Retrospective Study | 1 time point: 0-10 years post injury
  VOR time constant in response to a step rotation (initial 140°/s acceleration/deceleration and a 60°/s fixed-chair velocity) stimulus . Time constant (seconds) where a higher time constant is clinically better. Range 0-40s.
Patient reported outcome measure: Retrospective Study | 1 time point: 0-10 years post injury
  PROM (patient reported outcome measure) vertigo severity scale.15 questions rated 0-4. Score range =0-60 where lower scores indicate a better clinical outcome
Clinical measure of walking: Retrospective Study | 1 time point: 0-10 years post injury
  Dynamic Gait Assessment (DGA). Eight tasks scored 0-3. Total range = 0-24 with a higher score indicating better walking ability.
Clinical measure of balance: Retrospective Study | 1 time point: 0-10 years post injury
  Clinical measures of balance sharpened Romberg (tandem stance). The length of time a person is able to stand in the eyes open, tandem stance position is recorded up to a maximum of 30 seconds.
Posturography: Retrospective Study | 1 time point: 0-10 years post injury
  Postural sway quotient. Postural sway (mm/s) is measured via force plates. The ratio of the sway with eyes open and eyes closed is calculated (unitless ratio).
Perception of verticality: Retrospective Study | 1 time point: 0-10 years post injury
  Rod and Disk test: The ability to orientate a line to vertical is assessed with / without visual distractors. The error from vertical is recorded in degrees. Outcomes range from 0-180 degrees where lower numbers indicate better verical perception.
Functional MRI response to an optokinetic stimulus: Retrospective Study | 1 time point: 0-10 years post injury
  Regions of interest will also assess changes in activation with an optokinetic stimulus compared to rest in cortical and subcortical sites that process vestibular information namely the insulo-parietal cortex and hippocampus and sites that process other sensory information namely the visual cortex and somatosensory cortex
Vestibular Evoked myogenic Potentials latency: Retrospective Study | 1 time point: 0-10 years post injury
  Galvanic and Auditory Vestibular Evoked myogenic Potentials (VEMPs) will be assessed and the latency of evoked responses measured in milliseconds.
Vestibular Evoked myogenic Potentials amplitude: Retrorospective Study | 1 time point: 0-10 years post injury
  Galvanic and Auditory Vestibular Evoked myogenic Potentials (VEMPs) will be assessed and the amplitude of evoked responses measured in millivolts.

IPD SHARING:
Plan to Share IPD: Yes
Following study completion and publication of results anonymous data sets of clinical and laboratory outcome measures will be made available to other research teams on written request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will become available on study completion and after publication of results.
Access Criteria: Access to data will be via written request from other relevant healthcare professionals and research groups.

REFERENCES:
- [Background] Gempp E, Louge P. Inner ear decompression sickness in scuba divers: a review of 115 cases. Eur Arch Otorhinolaryngol. 2013 May;270(6):1831-7. doi: 10.1007/s00405-012-2233-y. Epub 2012 Oct 26. PMID 23100085
- [Background] Tremolizzo L, Malpieri M, Ferrarese C, Appollonio I. Inner-ear decompression sickness: 'hubble-bubble' without brain trouble? Diving Hyperb Med. 2015 Jun;45(2):135-6. PMID 26165540
- [Background] Mitchell SJ, Doolette DJ. Pathophysiology of inner ear decompression sickness: potential role of the persistent foramen ovale. Diving Hyperb Med. 2015 Jun;45(2):105-10. PMID 26165533
- [Background] Landolt JP, Money KE, Topliff ED, Ackles KN, Johnson WH. Induced vestibular dysfunction in squirrel monkeys during rapid decompression. Acta Otolaryngol. 1980;90(1-2):125-9. doi: 10.3109/00016488009131707. PMID 6969520
- [Background] Landolt JP, Money KE, Topliff ED, Nicholas AD, Laufer J, Johnson WH. Pathophysiology of inner ear dysfunction in the squirrel monkey in rapid decompression. J Appl Physiol Respir Environ Exerc Physiol. 1980 Dec;49(6):1070-82. doi: 10.1152/jappl.1980.49.6.1070. PMID 6969248
- [Background] Kurata N, Kawashima Y, Ito T, Fujikawa T, Nishio A, Honda K, Kanai Y, Terasaki M, Endo I, Tsutsumi T. Advanced Magnetic Resonance Imaging Sheds Light on the Distinct Pathophysiology of Various Types of Acute Sensorineural Hearing Loss. Otol Neurotol. 2023 Aug 1;44(7):656-663. doi: 10.1097/MAO.0000000000003930. Epub 2023 Jun 29. PMID 37400150
- [Background] Song CI, Pogson JM, Andresen NS, Ward BK. MRI With Gadolinium as a Measure of Blood-Labyrinth Barrier Integrity in Patients With Inner Ear Symptoms: A Scoping Review. Front Neurol. 2021 May 20;12:662264. doi: 10.3389/fneur.2021.662264. eCollection 2021. PMID 34093410
- [Background] Vargas-Figueroa VM, Caceres-Chacon M, Labat EJ. Scuba Diving-Induced Inner-Ear Pathology: Imaging Findings of Superior Semicircular Canal and Tegmen Tympani Dehiscence. Am J Case Rep. 2024 Jan 2;25:e941558. doi: 10.12659/AJCR.941558. PMID 38163945
- [Background] Gempp E, Louge P, de Maistre S, Morvan JB, Vallee N, Blatteau JE. Initial Severity Scoring and Residual Deficit in Scuba Divers with Inner Ear Decompression Sickness. Aerosp Med Hum Perform. 2016 Aug;87(8):735-9. doi: 10.3357/AMHP.4535.2016. PMID 27634609
- [Background] Curthoys IS, Halmagyi GM. Vestibular compensation: a review of the oculomotor, neural, and clinical consequences of unilateral vestibular loss. J Vestib Res. 1995 Mar-Apr;5(2):67-107. PMID 7743004
- [Background] McDonnell MN, Hillier SL. Vestibular rehabilitation for unilateral peripheral vestibular dysfunction. Cochrane Database Syst Rev. 2015 Jan 13;1(1):CD005397. doi: 10.1002/14651858.CD005397.pub4. PMID 25581507
- [Background] Darlington CL, Smith PF. Molecular mechanisms of recovery from vestibular damage in mammals: recent advances. Prog Neurobiol. 2000 Oct;62(3):313-25. doi: 10.1016/s0301-0082(00)00002-2. PMID 10840152
- [Background] Bense S, Bartenstein P, Lochmann M, Schlindwein P, Brandt T, Dieterich M. Metabolic changes in vestibular and visual cortices in acute vestibular neuritis. Ann Neurol. 2004 Nov;56(5):624-30. doi: 10.1002/ana.20244. PMID 15449325
- [Background] Hong SK, Kim JH, Kim HJ, Lee HJ. Changes in the gray matter volume during compensation after vestibular neuritis: a longitudinal VBM study. Restor Neurol Neurosci. 2014;32(5):663-73. doi: 10.3233/RNN-140405. PMID 25096973
- [Background] Helmchen C, Klinkenstein J, Machner B, Rambold H, Mohr C, Sander T. Structural changes in the human brain following vestibular neuritis indicate central vestibular compensation. Ann N Y Acad Sci. 2009 May;1164:104-15. doi: 10.1111/j.1749-6632.2008.03745.x. PMID 19645887